CLINICAL TRIAL: NCT06207864
Title: Participant Engagement - Cancer Genome Sequencing (PE-CGS) Research Center: Engagement of American Indians of Southwestern Tribal Nations in Cancer Genome Sequencing
Brief Title: Engagement of American Indians of Southwestern Tribal Nations in Cancer Genome Sequencing
Acronym: PE-CGS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: INST 2108; NCI-2023-02462 (Other: NCI); 5U2CCA252973 (NIH)
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-05

CONDITIONS: Malignant Neoplasm
Keywords: PE-CGS; Southwestern Tribal Nations; Cancer Genome Sequencing; American Indians
MeSH Terms: conditions — Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Category 1 (biospecimens, surveys, interviews) (Experimental): Cancer patients and survivors undergo collection of tissue, blood, saliva, and stool samples on study for genomic sequencing and microbiome analysis. Cancer patients and survivors also complete surveys and interviews on study pre and post intervention.
  Interventions: Procedure: Biospecimen Collection; Procedure: Return of Results; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of tissue, blood, saliva, and stool samples
  Other Names: Biological Sample Collection; Specimen Collection
Procedure: Return of Results — Receive results
Other: Survey Administration — Surveys and Interviews

SUMMARY:
This clinical trial studies engagement strategies for recruiting American Indians (AI) of Southwestern Tribal Nations for cancer genome sequencing. American Indians in the Southwest have higher rates of some types of cancer, such as cancers that arise in the liver, kidney, breast, and colon. American Indians with cancer may also live for less time than people from other population groups who have been treated for the same cancer. Damage to the cells of the body, acquired as people live, grow older, and are exposed to the environment, causes genetic changes in cells that can lead to cancer. This study may help researchers learn how these genetic changes in cells cause cancer and understand how and why cancer is arising in American Indians in the Southwest. This may help better prevent and treat cancer in the future.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

The overall objective of the PE-CGS Research Center is to develop culturally appropriate, respectful, trusted, and collaborative means to engage and recruit American Indians affected by cancer (newly diagnosed cancer patients, patients undergoing cancer treatment, and cancer survivors) for molecular characterization of their tumors.

The clinical trial is embedded in the Patient Engagement Unit (PEU) jointly with the Engagement Optimization Unit (EOU)

The specific objectives for the PEU are to:

1. Conduct direct participant engagement with cancer patients/survivors, community advisors, and partners to refine and optimize methods/processes;
2. Identify, recruit and consent eligible AI cancer patients/survivors;
3. Implement tissue acquisition, epidemiologic, behavioral, and clinical data collection, conduct continuous assessment of performance benchmarks;
4. Return clinical grade and clinically useful genomic data to participants with navigation to counseling and clinical resources as warranted and as they select.

The specific objectives of the EUO are to:

1. Finalize consenting process and informed consent by direct engagement of AI cancer patients, survivors, healthcare providers, genetic counselors, consenting staff, tribal and spiritual leaders and tribal governance;
2. Determine AI cancer patients' and survivors' knowledge, attitudes, cultural beliefs, information needs, and communication preferences and practices regarding clinical genomics testing;
3. Determine AI cancer patients' and survivors' perspectives on strategies to engage and recruit participants for clinical genomics testing.

ELIGIBILITY:
Inclusion Criteria:

* The PE-CGS Research Center is only recruiting and sequencing tumors for adult-onset cancers (patients and survivors) among the American Indian Tribes, Nations, and Pueblos of New Mexico and adjacent states
* Male or female adults (18 years) or older
* Cancer patient undergoing active treatment or a cancer survivor
* Self-identify as American Indian

Exclusion Criteria:

* Cognitively impaired
* Adults unable to consent for themselves
* Individuals who are not yet adults
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1001 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Enrolled Participants | Up to 18 months
  Number and percent of eligible participants enrolled and consented
Data participation rate | Up to 18 months
  Number and percent of eligible participants who complete, or partially complete, baseline and follow up data collection of epidemiological assessments and follow up data collection of epidemiological assessments
Biospecimen participation rate | Up to 18 months
  Number and percent of enrolled participants for whom biospecimens are collected and processed for genomic analysis
Rate of comprehensive genomic analysis completion | Up to 18 months
  Number and percent of participants/samples that undergo successful comprehensive genomic and bioinformatic analysis
Rate of successful return of clinical genetic/genomic results | Up to 18 months
  Number and percent of participants who elect to receive clinical genetic/genomic results and incidental findings
Rate of new threptic intervention as a result of participation | Up to 18 months
  Number and percent of participants/patients whose clinical genomic data facilitates therapeutic intervention
Rate of Preparatory and Optimization Phase completion | Up to 18 months
  Successful completion of the Preparatory and Optimization Phases

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Willman, MD, Principal Investigator — University of New Mexico Comprehensive Cancer Center; Nicole Hamblet, Study Director — University of New Mexico Comprehensive Cancer Center; Andrew Sussman, PhD, Study Director — University of New Mexico Comprehensive Cancer Center
Locations (1):
- University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] White MC, Espey DK, Swan J, Wiggins CL, Eheman C, Kaur JS. Disparities in cancer mortality and incidence among American Indians and Alaska Natives in the United States. Am J Public Health. 2014 Jun;104 Suppl 3(Suppl 3):S377-87. doi: 10.2105/AJPH.2013.301673. Epub 2014 Apr 22. PMID 24754660
- [Background] Jemal A, Ward EM, Johnson CJ, Cronin KA, Ma J, Ryerson B, Mariotto A, Lake AJ, Wilson R, Sherman RL, Anderson RN, Henley SJ, Kohler BA, Penberthy L, Feuer EJ, Weir HK. Annual Report to the Nation on the Status of Cancer, 1975-2014, Featuring Survival. J Natl Cancer Inst. 2017 Sep 1;109(9):djx030. doi: 10.1093/jnci/djx030. PMID 28376154
- [Background] Islami F, Miller KD, Siegel RL, Fedewa SA, Ward EM, Jemal A. Disparities in liver cancer occurrence in the United States by race/ethnicity and state. CA Cancer J Clin. 2017 Jul 8;67(4):273-289. doi: 10.3322/caac.21402. Epub 2017 Jun 6. PMID 28586094
- [Background] Ryerson AB, Eheman CR, Altekruse SF, Ward JW, Jemal A, Sherman RL, Henley SJ, Holtzman D, Lake A, Noone AM, Anderson RN, Ma J, Ly KN, Cronin KA, Penberthy L, Kohler BA. Annual Report to the Nation on the Status of Cancer, 1975-2012, featuring the increasing incidence of liver cancer. Cancer. 2016 May 1;122(9):1312-37. doi: 10.1002/cncr.29936. Epub 2016 Mar 9. PMID 26959385
- [Background] Nir I, Wiggins CL, Morris K, Rajput A. Diversification and trends in biliary tree cancer among the three major ethnic groups in the state of New Mexico. Am J Surg. 2012 Mar;203(3):361-5; discussion 365. doi: 10.1016/j.amjsurg.2011.12.002. Epub 2012 Jan 10. PMID 22236535
- [Background] Melkonian SC, Jim MA, Haverkamp D, Wiggins CL, McCollum J, White MC, Kaur JS, Espey DK. Disparities in Cancer Incidence and Trends among American Indians and Alaska Natives in the United States, 2010-2015. Cancer Epidemiol Biomarkers Prev. 2019 Oct;28(10):1604-1611. doi: 10.1158/1055-9965.EPI-19-0288. PMID 31575554
- [Background] Li J, Weir HK, Jim MA, King SM, Wilson R, Master VA. Kidney cancer incidence and mortality among American Indians and Alaska Natives in the United States, 1990-2009. Am J Public Health. 2014 Jun;104 Suppl 3(Suppl 3):S396-403. doi: 10.2105/AJPH.2013.301616. Epub 2014 Apr 22. PMID 24754655
- [Background] Hoffman RM, Espey DK, Rhyne RL, Gonzales M, Rajput A, Mishra SI, Stone SN, Wiggins CL. Colorectal cancer incidence and mortality disparities in new Mexico. J Cancer Epidemiol. 2014;2014:239619. doi: 10.1155/2014/239619. Epub 2014 Jan 2. PMID 24527035
- [Background] Sauer AG, Siegel RL, Jemal A, Fedewa SA. Updated Review of Prevalence of Major Risk Factors and Use of Screening Tests for Cancer in the United States. Cancer Epidemiol Biomarkers Prev. 2017 Aug;26(8):1192-1208. doi: 10.1158/1055-9965.EPI-17-0219. Epub 2017 May 17. PMID 28515109